CLINICAL TRIAL: NCT03575637
Title: Olanzapine Improves the Chemotherapy Tolerance of Advanced Gastric Cancer: a Prospective Randomized Controlled Phase II Clinical Study
Brief Title: Olanzapine Improves the Chemotherapy Tolerance of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Department of Gastrointestinal oncology, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Olanzapine
Record Dates: First submitted 2018-06-09; First posted 2018-07-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
Keywords: Olanzapine; Gastric Cancer; Tolerance
MeSH Terms: conditions — Stomach Neoplasms | interventions — Olanzapine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine intervention group (Experimental): Patients who have failed first-line treatment of advanced gastric cancer receive second-line treatment with paclitaxel regimen and olanzapine 5 mg QD.
  Interventions: Drug: Olanzapine
- Control group (No Intervention): Patients who have failed first-line treatment of advanced gastric cancer receive second-line treatment with paclitaxel regimen.

INTERVENTIONS:
Drug: Olanzapine — Patients who have failed first-line treatment of advanced gastric cancer receive second-line treatment with paclitaxel regimen and olanzapine 5 mg QD.
  Arms: Olanzapine intervention group

SUMMARY:
To explore whether adding olanzapine to paclitaxel chemotherapy could improve chemotherapy tolerance and improve patient quality of life and prolong treatment failure time (TTF) in advanced gastric cancer after failure of first-line chemotherapy.

This is a multi-center prospective randomized controlled open clinical study. Patients will formally be enrolled after they had been screened and signed informed consent. Baseline examinations will be started after entry into the group. Those who meet the criteria for inclusion and exclusion were dynamically randomized at 1: 1. The experimental group will receive olanzapine and paclitaxel until treatment failure and the control group will receive paclitaxel until treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent;
2. Age more than 18 years of age;
3. Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction;
4. Locally advanced recurrent or metastatic disease;
5. Have received systemic first-line chemotherapy and confirmed first-line treatment failure (platinum combined with fluorouracils);
6. Subjects' baseline blood routine and biochemical indicators meet the following criteria Hemoglobin ≥90g/L The absolute neutrophil count (ANC) is ≥1.5×10^9/L. Platelets ≥100×10^9/L ALT, AST ≤ 2.5 times the normal upper limit, ≤ 5 times the normal upper limit (with liver metastasis) ALP≤2.5 times normal upper limit, ≤ 5 times normal upper limit (with liver or bone metastases) Serum total bilirubin <1.5 times normal upper limit Serum creatinine <1.5 times normal upper limit Serum albumin ≥30g/L
7. KPS score ≥ 60 points;
8. Life expectancy ≥ 3 months.

Exclusion Criteria:

1. Does not meet the above selection criteria;
2. The first-line treatment uses paclitaxel-based drugs;
3. Pregnancy and lactation women;
4. Allergies to research drugs or people with metabolic disorders;
5. History of organ transplantation (including bone marrow autologous transplantation and peripheral stem cell transplantation);
6. Those who have been receiving systemic steroids for a long period of time (Note: Short-term users may be discontinued >2 weeks for inclusion);
7. Brain metastasis;
8. With severe infections need treatment;
9. Accompanied by dysphagia active peptic ulcer complete or incomplete intestinal obstruction active gastrointestinal bleeding perforation etc;
10. Severe liver diseases (such as liver cirrhosis etc.) kidney disease respiratory diseases or chronic diseases such as diabetes high blood pressure that cannot be controlled;
11. Having other malignant tumors within 5 years except non-melanoma skin cancer and cervical cancer in situ;
12. Heart disease with markedly abnormal electrocardiogram or clinical symptoms such as congestive heart failure marked coronary heart disease uncontrolled arrhythmia high blood pressure or previous myocardial infarction within 12 months or cardiac function Class III or IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
time to treatment failure | 2 year
  From randomization to exit the trial, the reasons for withdrawal may be patients' refusal, disease progression, patient death, and adverse events etc.

SECONDARY OUTCOMES:
side effect | 2 years
  Incidence of nausea and vomiting; Weight change; Drug exposure; Drug cumulative dose.
Progression free survival time (PFS), overall survival time (OS). | 2 years
  Progression free survival time (PFS), overall survival time (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No